CLINICAL TRIAL: NCT03009734
Title: A Prospective, Single Center, Randomized, Double-blind, Placebo Controlled Study in Two Phases to Evaluate the Safety and Efficacy of ATx201 as a Topical Antibiotic Agent
Brief Title: Evaluation of ATx201 as a Topical Antibiotic Agent
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DECOLAD
Record Dates: First submitted 2016-12-22; First posted 2017-01-04 (Estimated); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Infection, Bacterial
MeSH Terms: conditions — Bacterial Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ATx201 (2% dermal formulation A) and Placebo (Other)
  Interventions: Drug: ATx201 dermal formulations 2%
- ATx201 (2% dermal formulation B) and Placebo (Other)
  Interventions: Drug: ATx201 dermal formulations 2%
- ATx201 (2% dermal formulation C) and Placebo (Other)
  Interventions: Drug: ATx201 dermal formulations 2%

INTERVENTIONS:
Drug: ATx201 dermal formulations 2% — Topical application of ATx201 dermal formulations 2%

SUMMARY:
AntibioTx is developping ATx201 as a topical product for treatment of skin infections, including infected atopic dermatitis.

DETAILED DESCRIPTION:
Treatment of skin infections, including infected atopic dermatitis, is plagued by inactivity of or resistance towards the main topical antibiotics. Accordingly, the infections are either not effectively treated or harsher systemic antibiotics with side effects are needed.

Infections in atopic dermatitis are predominantly caused by Staphylococcus aureus and various species of Streptococcus. ATx201 is a potent antibiotic against these and other organisms. ATx201 overcomes current resistance problems such as methicillin resistant Staphylococcus aureus (MRSA), vancomycin resistant enterococci (VRE) as well as resistance towards all topical antibiotics. ATx201 also exhibits an extraordinarily strong ability to delay the onset of de novo resistance compared to currently marketed antibiotics.

The study is a combined Phase I/II study with 36 healthy volunteers and 40 patients.

The primary objective is to demonstrate the safety and tolerability of new topical formulations of ATx201 in healthy volunteers, and in a population of patients with infected atopic dermatitis. Efficacy of ATx201 in eradicating S. aureus compared to vehicle after 4 and 7 days of treatment will be evaluated. In Phase I of the study, three formulations of ATx201 including the respective Placebos will be applied to healthy volunteers. One formulation will advance into Phase II, where patients will be treated with the respective formulation or Placebo.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria:

* Signed and dated informed consent has been obtained
* Age 18 - 70 years
* Male or female
* Female subjects of childbearing potential must be confirmed not pregnant by a negative urine pregnancy test prior trial treatment
* Female subjects of childbearing potential must be willing to use effective contraceptive at trial entry until completion
* Male subjects must agree to use adequate contraception for the duration of the trial

Additional inclusion criteria for Phase II of the study:

* Localized disease (e.g. flexural eczema in a more or less symmetrical distribution on arms) where two individual lesions each covering an area between 10-200 cm2 and where each individual lesion has an investigators global assessment score between 1-3.
* Additional localized lesion of area between 10-200 cm2 and where the individual lesion has an investigators global assessment score between 1-3.
* Total localized disease not exceeding 20 % body surface area
* Colonization of lesions with S.aureus as determined by cultivation

General exclusion criteria

* Clinically relevant abnormalities in the laboratory testing, vital signs, ECG ( Phase I only) or physical examination
* Presence of any skin condition (scars, tattoos,…) that would interfere with the placement of study medication
* History of irritation to topical products
* Current acute or chronic disease unless considered clinically irrelevant by the Investigator
* Relevant history of malignancy, of renal, hepatic, cardiovascular, respiratory, gastrointestinal, musculoskeletal, skin (particularly at the site of drug application), haematological, endocrine or neurological diseases that may interfere with the aim of the study
* Positive HIV serology or evidence of active hepatitis
* Ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients of the study drugs (test, reference)
* History of drug or alcohol abuse (>2 drinks/day, defined according to USDA Dietary Guidelines 2005)
* caffeine (>5 cups coffee/tea/day) or tobacco abuse (consumption of 5 or more cigarettes/week)
* abnormal or special diet (e.g. vegetarian diet)
* Blood donations during 6 weeks prior to this study or planned within 6 weeks after the last blood withdrawal
* Subject considered unable or unlikely (per Investigator judgment) to comply with safety and PK profiling requirements (follow-up visits)
* Subjects who are pregnant (as determined by a positive pregnancy test at the screening visit) or lactating
* Participation in another clinical trial with an investigational day within 4 weeks before screening

Additional exclusion criteria for Phase I of the study:

* Regular use of medications
* Use of any dermatological drug therapy on the arms within 14 days before day 1 of this study

Additional exclusion criteria for Phase II of the study:

* Treatment with antibiotics (systemic or topical) within the past 3 months and during the study
* Treatment with drugs that affect the immune system within the past 3 months and during the study
* Treatment with topical steroids and calcineurin inhibitors 1 week before and during the study treatment period
* Treatment with systemic steroids within the past month and during the study
* Use of disinfectant soaps within 1 week before screening and during the study treatment period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2016-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of new topical formulations of ATx201 | 7 days
  Number of subjects with treatment related adverse events. AEs will be classified into standardised terminology from the verbatim description (Investigator term) according to the MedDRA Coding Dictionary. AEs will be classified by MedDRA term and associated system organ class.
  The number and percentage of subjects reporting AEs will be summarised by treatment group, system organ class, MedDRA term, and Phase.

SECONDARY OUTCOMES:
Assessment of the impact of ATx201 on the treated atopic dermatitis lesion. To determine the systemic exposure of ATx201. | 4 and 7 days
  Will be assessed by the investigators global assessment (IGA score):
  0: Clear (no inflammatory signs)
  1. Almost clear (just perceptible erythema, just perceptible papulation/infiltration)
  2. Mild disease (mild erythema and mild papulation/infiltration)
  3. Moderate disease (moderate erythema, moderate papulation/infiltration)
  4. Severe disease (severe erythema, severe population/infiltration)
Treatment success, defined as a 100-fold reduction in the S. aureus colony count / cm2 of sampled skin lesion | 4 and 7 days
Local dermal tolerability at the sites of application | 7 days
  Will be assessed using the following dermal assessment score:
  0 = no evidence of irritation,
  1. = minimal erythema, barely perceptible,
  2. = definite erythema, readily visible; minimal edema or minimal papular response,
  3. = erythema and papule,
  4. = definite edema,
  5. = erythema, edema, and papule,
  6. = vesicular eruption,
  7. = strong reaction spreading beyond test site.
Safety and tolerability of new topical formulations of ATx201 | 4 and 15 days
  Number of subjects with treatment related adverse events. AEs will be classified into standardised terminology from the verbatim description (Investigator term) according to the MedDRA Coding Dictionary. AEs will be classified by MedDRA term and associated system organ class.
  The number and percentage of subjects reporting AEs will be summarised by treatment group, system organ class, MedDRA term, and Phase.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Zeitlinger, MD, Principal Investigator — General Hospital Vienna
Locations (1):
- Department of Clinical Pharmacology, General Hospital of Vienna, Vienna, Austria